CLINICAL TRIAL: NCT05750108
Title: Transcutaneous Vagal Nerve Stimulation to Prevent Tachyarrhythmias in Patients Early Following Myocardial Infarction: A Randomized Clinical Trial
Brief Title: Transcutaneous Vagal Nerve Stimulation to Prevent Tachyarrhythmias in Patients Early Following Myocardial Infarction
Acronym: EARLY-VAGUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Principal Investigator, Senior cardiology expert. Prof. Konstantinos P. Tsioufis, MD, PhD, FESC, FACC, Professor of Cardiology, Director of 1st Department of Cardiology, Hippokratio Hospital, University of Athens, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EARLY-VAGUS
Record Dates: First submitted 2023-01-30; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Myocardial Infarction; Tachyarrhythmia
Keywords: transcutaneous vagal nerve stimulation
MeSH Terms: conditions — Myocardial Infarction; Tachycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Transcutaneous Vagal Nerve Stimulation (Active Comparator)
  Interventions: Device: Parasym device (active, current (mA) < discomfort threshold)
- Sham Transcutaneous Vagal Nerve Stimulation (Sham Comparator)
  Interventions: Device: Parasym device (sham, current (mA) = 0)

INTERVENTIONS:
Device: Parasym device (active, current (mA) < discomfort threshold) — Active transcutaneous Vagal Nerve Stimulation (tVNS) (Parasym device, Parasym Health, Inc, London, UK) will be performed with a clip attached to the ear at 20 hertz (Hz), 250 microseconds (ms) at a current just below discomfort threshold for 30 minutes twice a day, starting on post-MI day 0. Stimulation will continue until 7 days post-MI or discharge.
  Arms: Active Transcutaneous Vagal Nerve Stimulation
Device: Parasym device (sham, current (mA) = 0) — Parasym device will be attached to the ear twice a day, turned on but current set to 0 milliamp (mA), starting on post-MI day 0. Stimulation will continue until 7 days post-MI or discharge.
  Arms: Sham Transcutaneous Vagal Nerve Stimulation

SUMMARY:
Among patients early following ST-segment (ST) elevation myocardial infarction, transcutaneous vagus nerve stimulation is associated with a reduce of the burden of premature ventricular contractions in the first 40 days post-myocardial infarction (MI).

The above hypothesis will be tested with a randomized, prospective, parallel, single-blind clinical trial. The expected study duration is approximately 12 months from the time the first subject is enrolled (planned for June 2023) to the time of study's termination date (December 2024). Patient enrollment is planned to take place at two major centers in Greece. The researchers will obtain approval by the institutional review board (IRB).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years
* ST-elevation myocardial infarction which is treated with a primary percutaneous coronary intervention
* Signed written informed consent by the patient for participation in the study and agreement to comply with the medication and the follow-up schedule

Exclusion Criteria:

A patient will be excluded from the study if one or more of all the following criteria are present:

* < 3 months after prior ablation
* Patients on amiodarone
* Patients with known thyroid issues, on renal-dialysis
* Life expectancy of < 12 months
* Complex congenital heart disease
* Cardiogenic shock
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal)
* Known channelopathy such as Brugada syndrome, long QT syndrome, or Catecholaminergic monomorphic ventricular tachycardia
* Symptomatic sinus bradycardia or sinus node dysfunction at baseline without an implantable pacemaker
* Complete heart block or trifascicular block without an implantable pacemaker
* Recurrent vasovagal syncope
* Pre-existing implantable cardioverter-defibrillator (ICD)
* Secondary prevention indication for an ICD (i.e. sustained ventricular arrhythmias occurring more than 48 hours after qualifying myocardial infarction (patients with ventricular arrhythmias occurring ≤48 hours of myocardial infarction, or with non-sustained ventricular tachycardia at any time, are not excluded))
* On the heart transplant list
* Recurrent unstable angina despite revascularisation (defined as ongoing chest pain or ischemic symptoms at rest or with minimal exertion despite adequate treatment with anti-anginal medications)
* Congestive heart failure New York Heart Association class IV, defined as shortness of breath at rest, which is refractory to medical treatment (not responding to treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of Ventricular tachycardia burden | 1, 7 and 40 days follow-up
  Patients will undergo noninvasive continuous ECG monitoring using a 24-hour Holter monitoring at 1, 7 and 40 days to evaluate their number of Premature ventricular contractions (PVCs) and number of Non-Sustain Ventricular Tachycardias (NSVT).

SECONDARY OUTCOMES:
Change of Heart Rate Variability | 1, 7 and 40 days follow-up
  Patients will undergo noninvasive continuous ECG monitoring using a 24-hour Holter monitoring at 1, 7 and 40 days to evaluate Heart Rate Variability
Change of Heart Rate Turbulence | 1, 7 and 40 days follow-up
  Patients will undergo noninvasive continuous ECG monitoring using a 24-hour Holter monitoring at 1, 7 and 40 days to evaluate Heart Rate Turbulence
Change of Deceleration Capacity (DC) | 1, 7 and 40 days follow-up
  Patients will undergo noninvasive continuous ECG monitoring using a 24-hour Holter monitoring at 1, 7 and 40 days to evaluate Deceleration Capacity
Change of Echocardiographic strain | 1, 7 and 40 days follow-up
  Patients will undergo echocardiography at 1, 7 and 40 days to assess Myocardial substrate lesions and Post-infraction fibrosis
Change of Left Ventricle Ejection Fraction (LVEF) | 1, 7 and 40 days follow-up
  Patients will undergo echocardiography at 1, 7 and 40 days to assess Left Ventricle Ejection Fraction
Change of Signal Averaged ECG | 1, 7 and 40 days follow-up
  Patients will undergo a 12-lead electrocardiogram at 1, 7 and 40 days
Change of T Wave alternans and equal indexes derived from holter monitoring | 1, 7 and 40 days follow-up
  Patients will undergo noninvasive continuous ECG monitoring using a 24-hour Holter monitoring at 1, 7 and 40 days
Change of QT duration | 1, 7 and 40 days follow-up
  Patients will undergo noninvasive continuous ECG monitoring using a 24-hour Holter monitoring at 1, 7 and 40 days
Pain assessment | 7 days follow-up
  Pain scores will be assessed on postoperative days 0-7 using the visual analog score (Scale 0-10). Zero for no pain and ten being the worst pain experienced. They will be obtained and recorded into the medical record by the nurse monitoring the subject as part of standard care
Number of participants with adverse effects | 7 days follow-up
  Number of participants with pruritus, flush, pain at the stimulation site

CONTACTS AND LOCATIONS:
Locations (4):
- Heart Rhythm Institute, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States
- Greece (2):
  - First Department of Cardiology, Hippocration General Hospital, National and Kapodistrian University of Athens, Athens, Attica
  - Athens Heart Center Amarousion, Athens, Attica
- Biomedical Engineering, Khalifa University of Science and Technology, Abu Dhabi, United Arab Emirates